CLINICAL TRIAL: NCT03307525
Title: A Pilot Study Assessing the Correlation of Preoperative Sensory Testing and Genetic Polymorphisms With Acute and Persistent Postoperative Pain
Brief Title: Pain After Breast Surgery
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Society for Ambulatory Anesthesia (SAMBA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00026402
Record Dates: First submitted 2017-10-03; First posted 2017-10-11 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot observational study assessing various predictors for acute pain and persistent pain following breast surgery for cancer.

ELIGIBILITY:
Inclusion Criteria:

* English speaking undergoing elective breast cancer surgery

Exclusion Criteria:

* Patients with recurrent cancer, metastasis, and previous breast surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing elective breast cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2015-12-22 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Acute Pain | 72 hours after surgery
  Maximum pain score reported postoperatively

SECONDARY OUTCOMES:
Persistent Pain | More than 6 months after surgery
  pain score ≥ 3 or pain that impacts daily life as indicated by a score >0 on any of the 7 daily activity questions more than 6 months after surgery

REFERENCES:
- [Derived] Habib AS, Kertai MD, Cooter M, Greenup RA, Hwang S. Risk factors for severe acute pain and persistent pain after surgery for breast cancer: a prospective observational study. Reg Anesth Pain Med. 2019 Feb;44(2):192-199. doi: 10.1136/rapm-2018-000040. Epub 2019 Jan 5. PMID 30700614